CLINICAL TRIAL: NCT04803825
Title: The Feasibility of Heavy-slow Resistance Training, Radial Extracorporeal Shockwave Therapy (rESWT) and Information and Advice. The NOrwegian Tennis Elbow (NOTE) Study
Brief Title: The NOrwegian Tennis Elbow (NOTE) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Håkon Sveinall, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109547
Record Dates: First submitted 2021-02-16; First posted 2021-03-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Lateral Epicondylitis; Tennis Elbow; Tendinopathy, Elbow
Keywords: Extracorporeal shock wave therapy; Heavy slow resistance exercise; Strength exercises
MeSH Terms: conditions — Tennis Elbow; Elbow Tendinopathy | interventions — Extracorporeal Shockwave Therapy; Counseling

STUDY DESIGN:
Intervention Model Description: The study is a prospective randomised controlled trial, feasibility trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heavy Slow Exercise (Experimental): One dedicated physiotherapist will supervise and instruct the exercise program on an individual basis. If the patient doesn't have access to a dumbbell, it will be offered free rental from the physiotherapy ward. Follow-up on the exercises will be scheduled as needed and tele rehabilitation will be offered as an option. Additionally to HSR exercises, participants will be instructed to perform daily stretches of the forearm.
  Interventions: Other: Heavy Slow Exercises
- Extracorporeal Shock wave therapy (Active Comparator): The patients will receive rESWT (SwissDolodClast/EMS) once a week for three sessions. The treatment will be given by a physiotherapist trained in using rESWT. The rESWT is given on the ECRB tendon insertion area.
  Interventions: Device: Extracorporeal Shock wave therapy
- Information and advice (Active Comparator): The information and advice group are given a single face-to-face session with a physiotherapist, lasting up to 60 minutes.
  Interventions: Other: Information and advice

INTERVENTIONS:
Other: Heavy Slow Exercises — * Load magnitude: A dumbbell as heavy as possible within the given repetitions and sets.
  * Number of repetitions: week 1: 15 reps, Week 2-3: 12 reps, Week 4-5: 10 reps, Week 6-8: 8 reps, Week 9-12: 6 reps
  * Number of sets: 3
  * Rest between sets: 2 - 3 min.
  * Number of exercise interventions: 2
  * Duration of experimental period: 12 weeks
  * Fractional and temporal distribution of the contraction modes per repetition and duration of one repetition: 3s concentric, 2s isometric: while change concentric/eccentric phase, 3s eccentric.
  * Rest in-between repetitions: No
  * Range of motion: Full range of motion
  * Intervention frequency: 3 times a week, with minimum 48 h recovery time in-between.
  Other Names: HSR
  Arms: Heavy Slow Exercise
Device: Extracorporeal Shock wave therapy — Two thousand impulses of shock waves are applied to the painful tendon, with a pressure between 1.5 and 3.0 bar (depending on what the patient tolerates). We use a power hand piece that provides energy of 0.01-0.35 mJ/mm2
  Other Names: rESWT
  Arms: Extracorporeal Shock wave therapy
Other: Information and advice — Information and advice are based on assessment and will comprise the standardized oral and written information. Participants will be educated regarding pain during and after activities and encouraged to be physically active. With only one session, there is great reliance on self-management. Thus, information and advice are made available through a handout.
  Arms: Information and advice

SUMMARY:
Trial Design:

The Norwegian Tennis Elbow (NOTE) study is a single-centre; three-armed, feasibility randomised controlled trial.

Aim:

The primary aim of this study is to pilot the methods proposed to conduct a definite RCT study.

Objectives:

* Measure the process of recruitment.
* Measure intervention adherence and acceptability.
* Measure outcome measure retention rate and completeness. The Patient-Rated Tennis Elbow Evaluation (PRTEE) will be used as the primary outcome measure.

Intervention:

Patients will be randomised to either: 1) Heavy slow resistance training (HSR), 2) Radial extracorporeal shock wave therapy (rESWT) or 3) Information and advice.

Follow-up will be after 3 and 6 months.

DETAILED DESCRIPTION:
Background:

Lateral epicondylalgia, also known as tennis elbow, cause functional disability with high costs due to productivity loss, healthcare use and sickness absence. Evidence shows that physiotherapy is the most preferred patient treatment among Norwegian patients. However, the most efficient treatment for chronic tennis elbow is yet to be acknowledged. Exercises are a commonly used modality for tennis elbows. However, contradictory to lower limb tendinopathies, a pragmatic heavy slow resistance (HSR) exercise training protocol for tennis elbow have not yet been investigated. Radial extracorporeal shock wave therapy (rESWT) is another widely used modality and evidence is spares and inconsistent, reviews conclude that more high quality studies are needed.

This feasibility study will provide methodological evidence that will play an important role in the development of future RCT. The project will include 60 patients with lateral epicondylalgia, these patients will be randomised to either: 1) HSR exercises 2) rESWT or 3) information and advice. The randomization sequence is computer-generated with blocks of variable size, which is unknown to the treater and the outcome assessor. A research assistant will supply the trial physiotherapist with allocations to which group. The investigator assessing the outcome measures will be blind to group allocation. Statistical analysis will be conducted on a blinded intention-to-treat basis. Due to the nature of the intervention in the study, blinding of the trial physiotherapist will not be possible.

Tele rehabilitation and welfare technology are rapidly increasing its usability and value. To investigate if tele rehabilitation is suitable for a RCT, the exercise group will be offered voluntary tele rehabilitation as an alternative to physical follow-up.

Aims:

The objectives that will be evaluate is; 1) the process of recruitment, 2) intervention adherence and acceptability and 3) the outcome measures.

1. The process of recruitment will be measured by descriptive statistics from the enrolment. If participants redraw after baseline testing or are unwilling to be randomized, the participant will be asked to describe the reason.
2. To measure adherence to the intervention, participants will be asked to fil out an exercise diary which will be controlled at follow up consultations and collected at 3 months. Usage of tele rehabilitation and percentage of participants meeting to their appointments will be measured with descriptive statistics after 3 months. The acceptability and understanding of the intervention will be measure by a -9/+9 likert scale for acceptability of treatment the second session after randomization and at 3 months.
3. The retention rate and completeness of data of the primary and secondary outcome measures for a future full power RCT will be measured with explorative outcomes.

Statistical plan:

The analysis will focus on descriptive statistics with confidence intervals for the variables obtained. The characteristics of the patients will be presented as means with SDs, as medians with IQR or as counts with percentages. Being a feasibility study, our main aim is to describe the study sample of patients with tennis elbow and to assess our ability to collect data. Hence, the investigators will not perform any imputation of missing data. Change in the main outcome from baseline to follow-up (3 and 6 months) will be analysed using generalised linear mixed models.

There will be performed studies evaluating the validity, reliability, interpretability and responsiveness of the The Patient-Rated Tennis Elbow Evaluation, maximum grip strength and pain free grip strength. To achieve adequate power for the evaluation of the psychometric properties of the outcome measures. 40 more tennis elbow participants receiving treatement as usal from our clinic will be added to these analysis, in addion to the 60 participants in the RCT.

Included participants will have an ultrasound examination of their elbow by a trained doctor at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Ability to fill in the questionnaires (understand oral and written Norwegian)
* Clinically diagnosed tennis elbow provoked by at least two of: Pain on pressure of the common extensor origin, Pain during power grip, Resisted wrist extension (Tomsen test), Resisted third finger extension (Maudsley´s test), Stretching of the extensors (Mill´s test)

Exclusion Criteria:

* Patients With significant Language issues (does not understand oral or written Norwegian
* Contraindications to ESWT (pregnancy, coagulation disturbance, connective tissues disease, epilepsy, use og pacemaker)
* Suspicion of other serious illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
The process of recruitment | 2 year
  Criteria for success is that >75 percent of patients should be eligible for randomization, >90% should be willing to be randomized, recruitment rate should be 3.75 participants per month.
Intervention adherence (appointments) | 3 months
  Criteria for success is that 90 percent meets to appointments (Either physically or tele)
Intervention adherence (training sessions) | 3 months
  In the HSR group ≥ 30 training sessions should be completed within 12 weeks,
Intervention acceptability and understandability | 3 months
  ≥ 10/20 within each group should rate the treatment ≥+3 "acceptable" and ≥ 10/20 within each intervention group should rate the treatment ≥+3 "understandable"
Retention and completeness of patient-reported outcome measures | 6 months
  The retention of completed patient-reported outcome measures (i.e. PRTEE, Quick DASH, EQ-5D-5L should be >75 percent.

SECONDARY OUTCOMES:
The Patient-Rated Tennis Elbow Evaluation (PRTEE) | 6 months
  The Patient-Rated Tennis Elbow Evaluation (PRTEE), formerly known as the Patient-Rated Forearm Evaluation Questionnaire (PRFEQ), is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis.The questionnaire is scored from 0 - 100 and a higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. Scores from The PRTEE questionaire will also be used calculate sample size in a future RCT.
Disabilities of the Arm, Shoulder and Hand Outcome Measure (Quick-DASH) | 6 months
  The Disabilities of the Arm, Shoulder and Hand Outcome Measure (Quick-DASH) questionnaire is an 11-item shortened version of the thirty-item DASH outcome measure. It measures physical function and symptoms related to upper-limb musculoskeletal disorders. The questionnaire is scored from 0 - 100 and a higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability.
The 5-level EQ-5D (EQ-5D-5L) | 6 months
  The 5-level EQ-5D (EQ-5D-5L) descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: Level 1: no problems, Level 2: slight problems, Level 3: moderate problems, Level 4: severe problems and Level 5: extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1 digit number that expresses the level selected for that dimension, The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A total of 3125 possible health states is defined in this way. For example state "12345" indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression.
The 5-level EQ-5D (EQ-5D-5L) VAS (EQ VAS) | 6 months
  The 5-level EQ-5D VAS (EQ VAS) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The EQ VAS is scored from 0 - 100 and a lower score indicate poorer health, higher scores indicate a better health. The EQ VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Pain free grip strength | 3 months
  Patients will hold a hand grip dynamometer (Jamar) in a standing position with a fully extended elbow in a neutral pronation/supination. The patient will be instructed to squeeze slowly and stop squeezing at the onset of pain; the values in kg will then be registered. The pain free grip strength is measured three times at the asymptomatic side, with a 20-second rest interval between each measurement and then the procedure is repeated at the symptomatic side. After tested in fully extended position the same procedure will be followed with a 90 degrees elbow flexion, and in a neutral pronation/supination.
Maximum grip strength | 3 months
  Patients will hold a hand grip dynamometer (Jamar) in a standing position with a fully extended elbow in a neutral pronation/supination. The patient will be instructed to squeeze with their maximum effort; the values in kg will then be registered. The maximum grip strength is measured three times at the asymptomatic side, with a 20-second rest interval between each measurement and then the procedure is repeated at the symptomatic side. After tested in fully extended position the same procedure will be followed with a 90 degrees elbow flexion, and in a neutral pronation/supination.
Maximum grip strength pain | 3 months
  Immediately after each of the 12 squeezes of maximum grip strength the physiotherapist will ask the patient to rate their pain on a 10 - point NRS scale where 0 indicate no pain and 10 the worst imaginable pain.
Global improvement | 3 months
  The Global improvement will measure the patients change from baseline. With a scale ranging from -5 to +5, where -5 is maximum worsening 0 is unchanged, and +5 is completely recovered. Patients will also answer whether they experience the change as meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Sveinall, PT, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researches who provide a methodologically sound proposal

REFERENCES:
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Macdermid J. Update: The Patient-rated Forearm Evaluation Questionnaire is now the Patient-rated Tennis Elbow Evaluation. J Hand Ther. 2005 Oct-Dec;18(4):407-10. doi: 10.1197/j.jht.2005.07.002. No abstract available. PMID 16271687
- [Background] Slade SC, Dionne CE, Underwood M, Buchbinder R. Consensus on Exercise Reporting Template (CERT): Explanation and Elaboration Statement. Br J Sports Med. 2016 Dec;50(23):1428-1437. doi: 10.1136/bjsports-2016-096651. Epub 2016 Oct 5. PMID 27707738
- [Background] Mokkink LB, Terwee CB, Patrick DL, Alonso J, Stratford PW, Knol DL, Bouter LM, de Vet HC. The COSMIN checklist for assessing the methodological quality of studies on measurement properties of health status measurement instruments: an international Delphi study. Qual Life Res. 2010 May;19(4):539-49. doi: 10.1007/s11136-010-9606-8. Epub 2010 Feb 19. PMID 20169472
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Derived] Sveinall H, Brox JI, Engebretsen KB, Hoksrud AF, Roe C, Johnsen MB. Heavy slow resistance training, radial extracorporeal shock wave therapy or advice for patients with tennis elbow in the Norwegian secondary care: a randomised controlled feasibility trial. BMJ Open. 2024 Dec 20;14(12):e085916. doi: 10.1136/bmjopen-2024-085916. PMID 39806585